CLINICAL TRIAL: NCT05938842
Title: Online DBT-Mindfulness Intervention for Symptoms in Multiple Sclerosis: Study Protocol of a Randomized Controlled Trial
Brief Title: Study Protocol of Online DBT-Mindfulness Intervention in Multiple Sclerosis
Acronym: ODMiMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Judit Bort, PhD in Welfare, Health and Quality of Life, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ODMiMS229/2022
Record Dates: First submitted 2023-06-22; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; online intervention; Dialectal behaviour therapy; Mindfulness
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: DBT is a modified version of cognitive-behavioural therapy that places additional emphasis on emotion regulation, distress tolerance, self-acceptance, and validation of experience, and consists in several types of interventions, including the skills training group. One of the module os DBT is Mindfulness, which practice the ability to observe thoughts and feeling as temporary, as opposed to reflections of the reality that are necessarily tru.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online DBT-Mindfulness intervention (Experimental): Experimental group Dialectical behavior therapy (DBT) is a type of cognitive behavioral intervention. The module of Mindfulness is directed to balance emotion with reasoning in order to achieve "wise mind", to act with awareness and to decrease characteristic mood dependent.
  Interventions: Behavioral: Online DBT-Mindfulness Intervention
- Online psychoeducational intervention (Active Comparator): Active control group,
  Interventions: Behavioral: Online psychoeducational intervention

INTERVENTIONS:
Behavioral: Online DBT-Mindfulness Intervention — The whole intervention exists of 10 sessions, one session a week for at least one hour and a half. The session 1 is tailored to address specific issues to people with MS, whereas the sessions 2 to 7 are based on DBT and mindfulness contents, and in sessions 7 to 10 introduced some contents of ACT. The program is based in teaching two different sets "what" and "how" (Linehan, 1993). The first skill "what", teaches patients to simply observe; in a second level, to describe, which implies the ability to put the name to what one has observed; and in the third, "what" skill patients learn to fully participate in their actions in the current moment and without self-consciousness (Soler et al., 2012). In the other hand, the skills of "how" are related to how observe, how to describe and how to participate. Moreover, some mindfulness skills such as "Observing the breath", "Half-smiling", "Awareness" are practice introduced as homework tasks.
  Arms: Online DBT-Mindfulness intervention
Behavioral: Online psychoeducational intervention — The active control group intervention will be based on a psycho-educational framework and will involve MS-related topics (Oz & Oz, 2020). The psychoeducational intervention will be conducted by a psychologist with experience in working with pwMS through group videoconference and will follow similar format as the DBT-Mindfulness intervention, except for the homework tasks. The participants will receive information about different aspects related to the disease (e.g., disease progression, disease-symptoms, stress management, nutrition, sleep hygiene, physical activity, social relationships). The content of the sessions of the psychoeducation program was created based on the current literature about MS. Similar psychoeducational programs were used in other studies before (Oz & Oz, 2020; Dowd et al., 2015).
  Arms: Online psychoeducational intervention

SUMMARY:
The goal of this clinical trial is to test an Online DBT-Mindfulness intervention in people with Multiple Sclerosis.

The results of the online DBT-Mindfulness intervention will be compared to an active control group (psychoeducational intervention) to see if they improve her emotion dysregulation and decentering, and consequently, this benefits also improve symptoms like anxiety, depression, distress, fatigue and quality of life in people with MS.

DETAILED DESCRIPTION:
Design The study design is a mixed-methods approach, under the concurrent nested design. Quantitative measures are the predominant method, therefore qualitative procedures will be hierarchically subsumed under quantitative procedures. The quantitative approach will serve to assess the effectiveness of a using online DBT-Mindfulness intervention to improve emotion dysregulation, and decentering in a randomized controlled trial (RCT), compared to an active control group (online psychoeducational intervention). In addition, qualitative measures will be used to complement and explain the results, and to know intervention usability and acceptability through the participant's experiences and perceptions.

Sample size In order to maximize participants' opportunities for interaction, peer support and practice skills; group size for each group must keep small (15-20 participants). Therefore, we will employ a convenience sample of 40 patients with MS. Estimating a loss of 20% of patients 48 patients will have to be recruited: 24 in the intervention and 24 in the control group.

Recruitment process Study recruitment will take place in outpatients of neurology diagnosed with MS at the Universitary Hospital of Vic (UHV). Firstly, project information will be disseminated at the neurology department of the UHV to recruit sample for the study. They will receive information regarding eligibility criteria and the recruitment protocol. Secondly, the neurologist will select potential participants that meet the inclusion and exclusion criteria and will create a list of those that willing to participate. Then, according to the procedures established by Ethics Committee of the UHV, the neurologist will contact the patients and ask for their consent to be contacted by telephone by the study researchers. Thirdly, participants who accepted will be invited for a face-to-face meeting. In this first encounter, participants will be provided with detailed information about the study (i.e. intervention characteristics, data collection, and risks and benefits of participating in the study). The participants will sign voluntarily the Informed Consent after reading and understanding the study information. In addition, it will be reminded that study participation is voluntary, and they will have the right to withdraw from the study at any time without disruption to their usual care.

Randomisation and allocation procedures Participants attending to the first face-to-face meeting will be provided with an identification code. Researchers will use an Excel file to create a random sequence of numbers allocating patients to the intervention and the active control group by a simple randomization process.

Blinding Both interventions will have similar look and structure of sessions, but different content whether the patient belongs to the intervention or active control group. The researcher, in charge of recording and monitoring data, will be blinded to the participant's group allocation. Due to the intervention is performed online, participants will be blinded if they will be receiving the DBT-Mindfulness or the psychoeducational treatment.

Intervention The interventions will be delivered in 1h-1h30 weekly sessions over a 10-week period via Zoom videoconferences. Adherence will be monitorised through attendance at the session schedule. Reminder emails previous to each sesssion will be used to improve adherence to interventions.

Online DBT-Mindfulness intervention DBT-Mindfulness intervention is an adaptation from the original DBT Skills Training Manual. The intervention was adjusted from the original program for patients with borderline personality disorder. In this intervention, mindfulness skills were taught in ten consecutive weeks and formal mindfulness practices were encouraged and reinforced. Modifications concerned information about MS and its psychosocial consequences and texts and examples applying to MS patients. The adaptation program was performed in collaboration with several experts (e.g., DBT experts, neurologist, neuropsychologist, researchers), through different online interviews.

The aim of the module of mindfulness is to balance emotion with reasoning in order to achieve "wise mind", to act with awareness and to decrease characteristic mood dependent. The whole intervention exists of 10 sessions, one session a week for at least one hour and a half. The session 1 is tailored to address specific issues to pwMS, whereas the sessions 2 to 7 are based on DBT and mindfulness contents, and in sessions 7 to 10 introduced some contents of ACT.

All group sessions will be facilitated by a clinical psychologist experienced in DBT intervention. Quality controls of the intervention will be carried out throughout the sessions, by means of video recordings that will be supervised by a psychologist certificated in DBT.

Online psychoeducational intervention The active control group intervention will be based on a psycho-educational framework and will involve MS-related topics. The psychoeducational intervention will be conducted by a psychologist with experience in working with pwMS through group videoconference and will follow similar format as the DBT-Mindfulness intervention, except for the homework tasks. The participants will receive information about different aspects related to the disease (e.g., disease progression, disease-symptoms, stress management, nutrition, sleep hygiene, physical activity, social relationships). The content of the sessions of the psychoeducation program was created based on the current literature about MS. Similar psychoeducational programs were used in other studies before.

Data collection Intervention effectiveness will be measured at baseline (T1: pre-group assignment), at the end of the intervention (T2: post-intervention, up to 10 week), and at three-months follow-up (T3: 3months). The baseline assessment will be realized in the first encounter with the patients in individual and face-to-face format. In this, the patients will complete the questionnaires with a specialist, that will last a maximum of 1h the assessment. Then at each time point, study participants will complete the same questionnaires in online format collected by researchers.

Data management The personal data of the individuals that participate at the project will we pseudoanonimised by the researcher and identifying information will not be shared with other participants of the project. Only the code assigned to participants in the study will be listed in the worklists. In the final report or in case of communicating these results to the scientific community, their identity will remain anonymous.

The monitorisation of quantitative data will be documented using a Research Electronic Data Capture (REDCap). REDCap is a secure web-based software System that allows researchers create online forms for data capture, management, and simple analysis. All the data uploaded to the REDCap will be anonymous.

Qualitative data will be collected by the research members (BM) at the end of the intervention (T2). Semi-structured interviews for qualitative data will be delivered face-to-face by one research members (BM), tape-recorded and transcribed verbatim. Overall data management will be done by the research members' staff at the University of Vic-Central University of Catalonia.

Data analysis Quantitative analysis Descriptive analysis will be provided for the primary and secondary outcomes, reporting the mean and standard deviation (SD). The homogeneity between groups at baseline will be validated using t-tests for independent samples, except in cases where the Mann-Whitney U-test is required as non-parametric alternatives, for each variable.

All randomized participants who undergo a baseline assessment will be included in the analysis, regardless of whether they drop out, withdraw, or are lost to follow-up during the study, in accordance with the intention-to-treat principle. The Shapiro-Wilk test will be used to assess the normality of quantitative variables.

The impact of the online DBT-Mindfulness against the psychoeducational intervention will be tested with mixed linear models with repeated measures. The analyses for primary (emotion dysregulation, decentering) and secondary outcomes (fatigue, depression, anxiety, stress, and quality of life) will be measured at the three assessment points,baseline (T1), postintervention (T2), and follow-up (T3). Covariance analyses will also be conducted, including age, gender, years of the disease, EDSS and MS type (only it there are more than one type of MS) and any differences between groups at baseline to provide a better estimate of the true effect of the intervention by assessing clinical significance.

Estimates of the size of treatment effects will be presented together with confidence intervals, in addition to significance tests (alpha level of 0.05). SPSS version 25.0 software will be used for statistical analyses.

Qualitative analysis Qualitative analysis will be performed with the Atlas.ti software. Semi-structurated interviews will be transcribed verbatim. Thematic analysis will be used to develop themes and categories in the qualitative data base according to: the feelings and thoughts related to the intervention, the satisfaction with the program and the care received by the professionals, and impeding and facilitator factors. We will conduct the analysisi of the transcripts in parallel with ongoing data collection. A researcher of the team (BM) will keep notes after each interview and throughout the analysis process. Initial codes will use vocabulary as close as possible to that use the participants themselves to avoid incorporating preconceptions into the analysis. Patient and professionals quotes to support the results will be identified and translated from Catalan/Spanish to English. Themes will be returned to all participants for verifcation. Credibility of the data will be achieved by reviewing the documents handwritten by the participants and using their complementary comments, as well as the prolonged commitment of the researcher with the data.

Ethical aspects The trial is developed according to the guidance of Good Clinical Practice established by the Comitè d'ètica de la UVic-UCC regarding its methodologic, ethical, and legal aspects. Moreover, if needed, ethics review and approval will be evaluated for all relevant aspects of the study by the CHV- Fores foundation committee prior the research initiation. The project will be carried out following the principles of the Declaration of Helsinki (2013-17), on medical research in people. The trial will be reported and patients that volunteer will be asked to sign a written informed consent prior to program participation. The confidentiality of the subjects will be in accordance with regulations of the Organic law of Protection of Personal Data 3/2018, of December 5, as well as the EU General Data Protection Regulation (2016/679, GDPR). In accordance with the Organic Law of 1/1982, of May 5, which protects the right to one's own image, empowers its owner to reproduce their own image and prohibits third parties from obtaining, reproducing and disclosing the person's image without their consent. Study results will be reported according to Consolidated Standards of Reporting Trials (CONSORT) recommendations and will also be reported in the ClinicalTrials.gov registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed MS by a neurologist
* to have internet access
* to have a Expanded Disability Status Scale (EDSS) score between 0-6'5
* to have adequate Catalan or Spanish language comprehension.

Exclusion Criteria:

* have a substantial cognitive dèficit
* be in concurrent individual or group psychotherapy
* have a history of schizophrenia or other psychotic symptoms
* have history of alcohol or substance abuse or dependence within 6 months of study entry
* have a substantial psychiatric disorder or met DSM 5 criteria for Major Depression or suicide ideation
* have meditation experience or are currently practicing meditation or yoga.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Changes in emotion dysregulation | baseline (pre-group assignment), at the end of the intervention (up to 10 weeks), and at three-months follow-up
  Changes in emotion dysregulation will be assessed by the 16-ítem Difficulties in Emotion Regulation Scale (DERS). Higher scores in this scale indicate greater emotion dysregulation (score range 16 to 80). The DERS has good internal consistency and test-retest reliability, and adequate convergent and discriminant validity in large community samples.
Changes in decentering | baseline (pre-group assignment), at the end of the intervention (up to 10 weeks) and at three-months follow-up
  Decentering will be measured using The Experiences Questionnaire (EQ), validated in the Spanish population. This instrument is a self - reported questionnaire that examine decentering and rumination. It showed a good reliability and it seems adequate to detect changes after mindfulness-based interventions.

SECONDARY OUTCOMES:
Changes in fatigue | Baseline (pre-group assignment), at the end of the intervention (up to 10 weeks), and at three-months follow-up
  The Modified Fatigue Impact Scale (MFIS) will be employed to assess fatigue severity. This questionnaire included 21 items and has been recommended by the Fatigue Guidelines Development Panel of the Multiple Sclerosis Council for Clinical Practice Guidelines. This scale was validated and demonstrated good psychometric properties in Spain.
Changes in depression and anxiety | Baseline (pre-group assignment), at the end of the intervention (up to 10 weeks), and at three-months follow-up
  The Hospital Anxiety and Depression Scale (HADS) is a 14- item measure of anxiety and depression symptoms during the previous week. The total score ranges from 0 to 42, and each subscale (HADS-Anxiety and HADS-Depression) includes 7 items with scores ranging from 0 to 21. Higher scores indicate higher symptom severity. The Spanish version has shown good psychometric properties and high internal consistency.
Changes in stress | Baseline (pre-group assignment), at the end of the intervention (up to 10 weeks), and at three-months follow-up (up to
  The Perceived Stress Scale (PSS-10) consists of 10 items which measure the degree to which a subject appraises situations as stressful during the last month. Scores range from 0 to 40, with higher scores reflecting higher perceived stress. The Spanish version has demonstrated adequate internal consistency, test-retest reliability, validity, and sensitivity to change.
Changes in QoL | Baseline (pre-group assignment), at the end of the intervention (up to 10 weeks), and at three-months follow-up
  QoL will be evaluated by the World Health Organization's WHOQOL-BREF quality of life assessment. The WHOQOL-BREF is a 26-item version of the WHOQOL-100 assessment and examined the individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. This scale has demonstrated good to excellent psychometric properties of reliability and performs well in preliminary tests of validity.

OTHER OUTCOMES:
Feasibility of the study | At the end of the intervention (up to 10 weeks)
  The feasibility of the programme (DBT-Mindfulness intervention) will be evaluated qualitatively in order to understand perceptions and experiences of the intervention participants. Individual semi-structured interviews will be performed. The interview schedule will consist of a series of broad, open-ended questions, and it will be structurized in three parts, exploring a) feelings and thoughts related to the intervention ; b) the satisfaction with the program and the care received by the professionals; and c) impeding and facilitator factors. Interviews will be performed until saturation of data achieved.

CONTACTS AND LOCATIONS:
Overall Officials: BRENDA MONTAÑÉS MASIAS, Principal Investigator — UVic-UCC
Locations (1):
- UVic-UCC, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soler J, Valdeperez A, Feliu-Soler A, Pascual JC, Portella MJ, Martin-Blanco A, Alvarez E, Perez V. Effects of the dialectical behavioral therapy-mindfulness module on attention in patients with borderline personality disorder. Behav Res Ther. 2012 Feb;50(2):150-7. doi: 10.1016/j.brat.2011.12.002. Epub 2011 Dec 14. PMID 22225697
- [Background] Soler J, Franquesa A, Feliu-Soler A, Cebolla A, Garcia-Campayo J, Tejedor R, Demarzo M, Banos R, Pascual JC, Portella MJ. Assessing decentering: validation, psychometric properties, and clinical usefulness of the Experiences Questionnaire in a Spanish sample. Behav Ther. 2014 Nov;45(6):863-71. doi: 10.1016/j.beth.2014.05.004. Epub 2014 Jun 2. PMID 25311294
- [Background] Feliu-Soler A, Pascual JC, Borras X, Portella MJ, Martin-Blanco A, Armario A, Alvarez E, Perez V, Soler J. Effects of dialectical behaviour therapy-mindfulness training on emotional reactivity in borderline personality disorder: preliminary results. Clin Psychol Psychother. 2014 Jul-Aug;21(4):363-70. doi: 10.1002/cpp.1837. Epub 2013 Mar 14. PMID 23494767
- [Background] Oz HS, Oz F. A psychoeducation program for stress management and psychosocial problems in multiple sclerosis. Niger J Clin Pract. 2020 Nov;23(11):1598-1606. doi: 10.4103/njcp.njcp_462_19. PMID 33221788